CLINICAL TRIAL: NCT02010268
Title: Evaluation of a Clinico-biological Predictive Score of Enterocolitis and Enteropathy of the Preterm Neonates. Usefulness of the Rapid Assay of the Faecal Calprotectin.
Brief Title: Use of Faecal Calprotectin to Predict Enteropathy of the Preterm Neonates
Acronym: CALPROPREMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P111104
Record Dates: First submitted 2013-08-02; First posted 2013-12-12 (Estimated); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Enteropathy, Necrotizing Enterocolitis
Keywords: Faecal calprotectin; Feces; Preterm neonates; Enterocolitis; Enteropathy; Necrotizing
MeSH Terms: conditions — Intestinal Diseases; Enterocolitis, Necrotizing; Enterocolitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- preterm neonates (Experimental): Preterm neonates (birth before 33 weeks of gestation)
  Interventions: Other: Collection of stool samples

INTERVENTIONS:
Other: Collection of stool samples — A stool sample will be collected once a week from birth until discharge from the hospital, and every day during digestive episodes, that is to say during an interruption of enteral nutrition for more than 48 hours.

SUMMARY:
This study aims to evaluate a clinico-biological predictive score, associating the faecal calprotectin, for the diagnosis of enterocolitis and enteropathy of the preterm neonates.

DETAILED DESCRIPTION:
Enteropathy and necrotizing enterocolitis (NEC) are digestive emergencies in premature neonates which represent a major concern for the vital prognosis. It is therefore important to propose a tool for early diagnosis of these intestinal complications in order to avoid extended interruptions of enteral feeding at a period of life where growth (and digestive maturation) is in the foreground. Currently, the diagnosis of digestive impairment is based on classical clinical, biological (CRP, procalcitonin, fecal calprotectin, NFS) and radiological (abdomen without preparation) approaches, which induce on one hand a prolonged interruption of enteral feeding sometimes useless and even harmful for the intestinal maturation and, secondly, the establishment of a parenteral nutrition which is not risk-free. The study propose to dose the fecal calprotectin, a non-invasive marker of digestive inflammation, in order to validate the threshold decision proposed in a pilot study (350 µg/g of feces). Measurement of fecal calprotectin levels will be used as an integrated tool to build a powerful screening score combined to the usual parameters used in routine care for the diagnosis of and enteropathy and necrotizing enterocolitis (NEC) in premature neonates. A cohort of preterm infants born at a gestational age of 33 weeks or less will be included from birth. A stool sample will be collected from the diaper once a week, from birth until discharge from the hospital, and every day during gastrointestinal events (interruption of enteral feeding over 48 hours). The study will evaluate the performance of the rapid assay of fecal calprotectin by quantitative immunochromatography compared to the reference method by enzyme-linked immunosorbent assay (ELISA).

ELIGIBILITY:
Inclusion Criteria:

* Infants prematurely born at a gestational age of 33 weeks or less (or before the 7th month of pregnancy).
* Patient whose parents or holders of parental authority signed an informed consent.

Exclusion Criteria:

* Patient with a malformation.
* Lack of signature of the consent by parents or holders of parental authority.

Max Age: 33 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 122 (Actual)
Dates: Start 2013-09-30 (Actual); Primary Completion 2015-02-22 (Actual); Study Completion 2015-02-22 (Actual)

PRIMARY OUTCOMES:
fecal calprotectin level | From birth to hospital discharge (3 months maximum).
  Quantification of fecal calprotectin in stool samples collected every week and the first 3 days during an interruption over 48 hours of enteral feeding

SECONDARY OUTCOMES:
Evaluation of the performance of fecal calprotectin rapid assay. | from birth to hospital discharge (3 months maximum)
  The measurement results of fecal calprotectin obtained by the rapid quantitative immunochromatography method, will be compared with those obtained by conventional reference method (ELISA).

CONTACTS AND LOCATIONS:
Overall Officials: Florence Campeotto, MD, PhD, Principal Investigator — Necker Hospital
Locations (1):
- Necker Hospital, Paris, France

REFERENCES:
- [Background] Campeotto F, Elie C, Rousseau C, Giuseppi A, Hachem T, Gobalakichenane P, Le Touzey M, de Stefano M, Butel MJ, Kapel N. Faecal calprotectin and gut microbiota do not predict enteropathy in very preterm infants. Acta Paediatr. 2021 Jan;110(1):109-116. doi: 10.1111/apa.15354. Epub 2020 Sep 1. PMID 32418251